CLINICAL TRIAL: NCT04522817
Title: CLBS119 (Autologous Peripheral Blood Derived CD34+ Cells) for Repair of COVID-19 Induced Pulmonary Damage
Brief Title: CLBS119 for Repair of COVID-19 Induced Pulmonary Damage
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Acute COVID-19 treatments have improved significantly leading to decreased use of ventilatory support. This, coupled with approval of a vaccine, has changed the profile/prognosis of patients and led to a lack of patients with long-term hypoxia.
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBS119-P01
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Covid-19
Keywords: Pneumonia; COVID; SARs-CoV-2; Pulmonary Inflammation; Respiratory Distress Syndrome; Lung Diseases; Lung Injury; Respiratory Tract Diseases; Respiratory Insufficiency; ARDS; pandemic; Corona Virus Infection; Coronavirus
MeSH Terms: conditions — COVID-19; Pneumonia; Respiratory Distress Syndrome; Lung Diseases; Lung Injury; Respiratory Tract Diseases; Respiratory Insufficiency; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLBS119 Active Treatment (Experimental): Single administration of CLBS119
  Interventions: Biological: CLBS119

INTERVENTIONS:
Biological: CLBS119 — Peripheral blood derived autologous CD34+ cells

SUMMARY:
This clinical trial will explore the safety and potential efficacy of CLBS119 for the repair of COVID-19 induced pulmonary damage in adults.

DETAILED DESCRIPTION:
This open-label clinical trial will explore the safety and potential efficacy of peripheral blood derived autologous CD34+ cells for the repair of COVID-19 induced pulmonary damage in adults. Eligible subjects will receive a single administration of CLBS119.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis with COVID-19 based on nasopharyngeal, oropharyngeal, or tracheobronchial aspirate SARS CoV-2 RT-PCR test
* Receiving or received ventilatory support for COVID-19 pneumonia/ARDS
* Evidence for ongoing pulmonary involvement based on P/F ratio <300
* Able to provide informed consent

Exclusion Criteria:

* Immunocompromised or current use of immunosuppressive agents other than corticosteroids
* History of autoimmune disease
* Evidence of multiorgan failure
* Subject is pregnant or lactating at the time of signing the consent
* Participation in any other clinical trial of an experimental treatment for COVID-19
* History of sickle cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through end of study (6 months)

SECONDARY OUTCOMES:
Change in oxygen saturation | Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Losordo, MD, Study Director — Chief Medical Officer, Caladrius Biosciences
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No